CLINICAL TRIAL: NCT05577143
Title: Evaluation of the Discriminatory Role of Blood TFPI-1 and TFPI-2 in Adult Colorectal Cancer
Brief Title: Blood Screening for Adult Colorectal Cancer
Acronym: BACCHUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021_0220; 2022-A00223-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer Colorectal
Keywords: Oncology; Biology
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group: All consecutive patients from participating centers with an abnormal colonoscopy (presence of mucosal lesions at endoscopy), with histological confirmation of colorectal cancer. These will be patients with one or more histologically confirmed adenocarcinomatous lesions (CRC+) located in the colonic frame or rectum, with or without synchronous liver metastases.
- Control group: All consecutive patients between 50 and 75 years of age for whom colonoscopy will be normal (no mucosal lesions). In this situation, histological examination is not performed.
- Polyp group: All consecutive patients for whom colonoscopy shows mucosal lesions that will be classified as polyps after histological examination.

SUMMARY:
Multicenter, inter-regional, case-control study with the primary objective of evaluating the discriminative power of the blood biomarker TFPI-1 to separate patients with histologically proven CRC from an asymptomatic control population between 50 and 75 years of age with normal colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected colorectal cancer for which colonoscopy is indicated.
* Patients between 50 and 75 years old, asymptomatic from the digestive point of view (for example referred for colonoscopy as part of a pre-operative check-up of an inguinal hernia or 3 months after an episode of complicated sigmoiditis), for whom a follow-up colonoscopy is indicated.

Note.

* If the post-inclusion colonoscopy is normal, no biopsy will be performed and patients will be assigned to the control group.
* If the colonoscopy performed after inclusion is abnormal (presence of at least one mucosal lesion), patients will be assigned to the "colorectal cancer" group or to the "polyps" group depending on the results of the anatomopathological analysis of the lesion(s)

Exclusion Criteria:

* All clinical situations outside of CRC that could increase TFPI-1 or 2 blood levels: acute coronary syndrome (unstable angina, acute myocardial infarction), severe sepsis, decompensated cirrhosis, pregnancy, chronic inflammatory bowel disease (Crohn's or ulcerative colitis), colitis or radiation rectitis.
* Endoscopic polypectomy without prior histological confirmation.
* Emergency (occlusion or peritonitis)
* Minor patients.
* Persons of full age under legal protection or unable to express their consent
* Persons not affiliated to a social security system or beneficiaries of such a system.
* Pregnant women, women in labor or nursing mothers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed up for colonoscopy in the gastroenterology and digestive surgery departments of 5 regional hospitals in northern France
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUC) of the TFPI-1 biomarker | At 2 months
  the AUC of the TFPI-1 biomarker to separate the 2 groups (CRC+ and control, i.e., asymptomatic population between 50 and 75 years with normal colonoscopy).

SECONDARY OUTCOMES:
AUC of the TFPI-2 biomarker to separate the 2 groups (CRC+ and control). | At 2 months
AUC of the discriminant score constructed by logistic regression with the 2 blood biomarkers as explanatory variables and the group type (CRC+ and control) as the variable to be explained. | At 2 months
Extension of c-index to the 3-group case proposed by Van Calster B et al. | At 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ZERBIB, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital HURIEZ - Chirurgie digestive et transplantation, Lille, France